CLINICAL TRIAL: NCT06517745
Title: Prone Positionning in Non Intubated ICU Patients With SARS-COV2
Brief Title: Effect of Prone Positionning in Non Intubated Patients
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of Anesthesiology and ICU department, Mongi Slim Hospital
Other Study IDs: COVID PP
Record Dates: First submitted 2024-07-22; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: SARS-CoV 2 Pneumonia; Acute Respiratory Distress Syndrome; Prone Positioning
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prone position group: Prone positioning sessions: at least 1 session per day session duration: at least 2 hours
  Interventions: Procedure: Prone positioning
- Control group: no prone positioning

INTERVENTIONS:
Procedure: Prone positioning — Prone positioning sessions: at least one session per day proning duration: 2 hours at least per session
  Groups: Prone position group

SUMMARY:
Retrospective single center study on the effect of awake prone positioning in ICU patients with severe hypoxemia related to SARS-COV2

DETAILED DESCRIPTION:
Retrospective, observational study on the effects of awake prone positioning on oxygenation, invasive mechanical ventilation requirement and mortality in non intubation patients with severe hypoxemia related to SARS-COV2 and regardeless of the oxygen supplementation method.

ELIGIBILITY:
Inclusion Criteria:

* All adult (> 18 years) patients, non intubated, with acute respiratory failure due to COVID-19 pulmonary infection

Exclusion Criteria:

* patients: hemodynamic instability and high doses of vasopressors
* patients with contraindications of prone positioning: pregnancy, recent abdominal surgery
* patients with pulmonay embolism
* patients requiring invasive mechanical ventilation for extra respiratory reasons: neurological failure, urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (> 18 years) patients admitted in the ICU:
  * with acute respiratory failure due to COVID-19 pulmonary infection
  * non intubated
  * regardeless of the exygenation method: HFONC, face mask, non invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Intubation | at day 7
  invasive mechanical ventilation requirement
Intubation | at day 14
  invasive mechanical ventilation requirement

SECONDARY OUTCOMES:
ICU mortality | at Day 14
  observed mortality rate in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided